CLINICAL TRIAL: NCT03396913
Title: Effectiveness of Intense Pulsed Light for Improving Signs and Symptoms of Dry Eye Disease Due to Meibomian Gland Dysfunction
Brief Title: Effectiveness of Intense Pulsed Light for Improving Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUM-VBU-M22-IPL-17-01
Record Dates: First submitted 2017-12-28; First posted 2018-01-11 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye Syndrome
Keywords: Intense Pulsed Light; Meibomian Gland Dysfunction; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to a study arm and a control arm. Subjects in the study arm will be treated with IPL and meibomian gland expression. Subjects in the control arm will be treated with sham and meibomian gland expression.
Who Masked: Participant
Masking Description: Subjects in the study arm will receive a series of IPL pulses using the M22 IPL handpiece. In subjects of the control arm, the device will be disabled. The subject will feel the lightguide on the skin, will hear clicking sounds, but no light will be actually produced by the M22 device. Since during treatment both eyes of the subject will be fully occluded, no subject will be able to see if the treatment is actual or sham. There is no way to completely mask the subjects, since the IPL generally causes slight redness of the skin, and in some patients is may also cause some discomfort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IPL followed by Meibomian Gland Expression (MGX) (Experimental): Subjects in the experimental arm with receive IPL followed by MGX: IPL pulses will be administered on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and below the lower eyelids. Following IPL therapy, subjects will undergo MGX of both eyelids in both eyes.
  Interventions: Device: IPL; Procedure: MGX
- Sham IPL followed by MGX (Sham Comparator): Subjects in the sham comparator arm with receive Sham IPL followed by MGX: Sham IPL pulses will be administered on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and below the lower eyelids. Following Sham IPL therapy, subjects will undergo MGX of both eyelids in both eyes.
  Interventions: Device: Sham IPL; Procedure: MGX

INTERVENTIONS:
Device: IPL — Intense pulsed light (IPL) is a non-invasive and non-laser light treatment that is FDA-approved for various conditions in dermatology. Subjects will receive a total of 4 IPL treatments over the course of the study, at intervals of 2 weeks. Each treatment will include applications of 10-15 IPL pulses in the malar region and close to the lower eyelids, followed by meibomian gland expression.
  Arms: IPL followed by Meibomian Gland Expression (MGX)
Device: Sham IPL — Sham intense pulsed light (IPL) will be implemented with an IPL device in which all light is blocked by a filter. Subjects will receive a total of 4 sham treatments over the course of the study, at intervals of 2 weeks. Each treatment will include applications of10-15 sham pulses in the malar region and close to the lower eyelids, followed by meibomian gland expression.
  Arms: Sham IPL followed by MGX
Procedure: MGX — Meibomian gland expression (MGX) will be implemented by squeezing the meibomian glands with the aid of two Q-tips positioned on either side of the meibomian glands, or with a meibomian gland expressor forceps

SUMMARY:
The aim of the current study is to examine the contribution of intense pulsed light (IPL) for relieving signs and symptoms of dry eye due to meibomian gland dysfunction. The effect of IPL will be examined in a study designed as a randomized controlled trial. In the study arm, subjects will undergo 4 treatment sessions, consisting of IPL pulses immediately followed by meibomian gland expression (MGX). In the control arm, subjects will undergo the same treatments, except that the IPL pulses will be disabled. For each subject, the duration of the study will be 10 weeks, as explained in the detailed description.

DETAILED DESCRIPTION:
Outcome measures (tear break-up time,meibography, self-assessed symptoms and close up photos of the lid margins) will be measured at baseline. All subjects will receive 4 treatments at 2 weeks intervals. In each treatment session, a subject allocated to the study group will be treated with intense pulsed light (IPL) administered in the malar region, from tragus to tragus including the nose, 2-3 mm below the lower eyelids. Immediately following the IPL administration, the subject will undergo meibomian gland expression (MGX) in both eyelids of both eyes. Subjects in the control arm will receive exactly the same treatment, except that the IPL administration will be sham. A single follow-up will occur at 10 weeks after the baseline (or 4 weeks after the 4th treatment session). At the follow-up, the changes in the outcome measures will be evaluated, and compared between the two arms.

For each subject, the duration of the study will be 10 weeks: 1st treatment at baseline; 2nd treatment at 2 weeks after baseline; 3rd treatment at 4 weeks after baseline; 4th treatment at 6 weeks after baseline; and a single follow-up at 10 weeks after baseline).

Statistically significant differences between the two arms will support the study hypothesis that IPL treatment itself provides relief to both signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand and sign an Informed Consent (IC) form
* 22-85 years of age
* Subject is able and willing to comply with the treatment/follow-up (FU) schedule and requirements
* In the study eye, Tear Breakup time (TBUT) ≤ 7 seconds
* In the study eye, Meibomian Gland Score (MGS) ≤ 12
* In the study eye, at least 5 non-atrophied meibomian glands in the lower eyelid
* Symptoms self-assessed using the Ocular Surface Disease Index (OSDI) questionnaire ≥ 23

Exclusion Criteria:

* Fitzpatrick skin type V or VI
* Contact lens wear within the month prior to screening
* Unwilling to discontinue use of contact lenses for the duration of the study
* Ocular surgery or eyelid surgery, within 6 months prior to screening
* Neuro-paralysis in the planned treatment area, within 6 months prior to screening
* Other uncontrolled eye disorders affecting the ocular surface, for example active allergies
* Current use of punctal plugs
* Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
* Uncontrolled infections or uncontrolled immunosuppressive diseases
* Subjects with ocular infections, within 6 months prior to screening
* Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 560 nm to 1200 nm, including: Herpes simplex 1 & 2, Systemic Lupus erythematosus, and porphyria
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Over exposure to sun, within 4 weeks prior to screening
* Use of prescription eye drops for dry eye, within 7 days prior to screening, excluding artificial tears and glaucoma drops
* Radiation therapy to the head or neck, within 12 months prior to screening
* Planned radiation therapy, within 8 weeks after the last treatment session
* Treatment with chemotherapeutic agent, within 8 weeks prior to screening
* Planned chemotherapy, within 8 weeks after the last treatment session
* New topical treatments within the area to be treated, or oral therapies, within 3 months prior to screening- except over-the-counter acetaminophen-based analgesics for pain management, new oral omega 3 fatty acid supplements and topical artificial tears
* Change in dosage of any systemic medication, within 3 months prior to screening
* Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period
* Legally blind in either eye
* History of migraines, seizures or epilepsy
* Facial IPL treatment, within 12 months prior to screening
* Any thermal treatment of the eyelids, including Lipiflow, within 6 months prior to screening
* Expression of the meibomian glands, within 6 months prior to screening
* In either eye, moderate to severe (Grade 3-4) inflammation of the conjunctiva, including: allergic, vernal or giant papillary conjunctivitis
* In either eye, severe (Grade 4) inflammation of the eyelid, including: blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy)
* Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, and severe ptosis
* Any systemic condition that may cause dry eye disease, including: Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, and Sjögren's syndrome
* Unwilling or unable to abstain from the use of medications known to cause dryness (e.g., isotretinoin, antihistamines) throughout the study duration. Subjects must discontinue these medications for at least 1 month prior to the baseline visit.
* Any condition revealed whereby the investigator deems the subject inappropriate for this study

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Dell, MD, Principal Investigator — Dell Laser Consultants; Rolando Toyos, MD, Principal Investigator — Toyos Clinic; Neel Desai, MD, Principal Investigator — The Eye Institute of West Florida
Locations (2):
- United States (2):
  - Toyos Clinic, Nashville, Tennessee
  - Dell Laser Consultants, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham+MGX: Sham IPL followed by meibomian gland expression (control group)
- IPL+MGX: Patients treated with IPL followed by meibomian gland expression (study group)
Period: Overall Study
Arm/Group | Sham+MGX | IPL+MGX
Started | 43 | 45
Completed | 43 | 39
Not Completed | 0 | 6
Not completed — Lost to Follow-up | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham+MGX | IPL+MGX | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.7) | 54.2 (14.3) | 55.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 10 | 25 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change of Baseline Tear Breakup Time (TBUT)
Description: Change of Tear breakup time (TBUT) in the study eye, from baseline to follow-up. TBUT is measured in seconds. Higher values mean better outcome.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Sham+MGX | IPL+MGX
Number analyzed (Participants) | 43 | 39
seconds | 0.75 (0.34) | 1.99 (0.36)

2. Secondary Outcome: Change From Baseline Ocular Surface Disease Index (OSDI)
Description: Change of self-assessed symptoms with the Ocular Surface Disease Index (OSDI) questionnaire, from baseline to follow-up. OSDI was collected per patient (one number per patient). The minimal number is 0 and the maximal number is 100. Higher scores mean worse outcome. A score of 0-12 is considered normal. A score of 13-22 is consistent with mild dry eye. A score of 23 to 32 is consistent with moderate dry eye. A score from 33 to 100 is consistent with severe dry eye.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham+MGX | IPL+MGX
Number analyzed (Participants) | 43 | 39
score on a scale | -25.9 (3.6) | -29.89 (3.78)

3. Secondary Outcome: Change From Baseline Eye Dryness Score (EDS)
Description: Change of self-assessed symptoms on a visual analog scale (VAS) , from baseline to follow-up, in both eyes. Values were collected separately for each eye. Correlation between eyes was removed by statistical methods. Scores were 0 (minimum) to 100 (maximum). Higher scores = worse outcome. VAS scores are not validated for dry eye. Hence, it is not known how to correlate VAS values to severity levels of dry eye. However, one can make estimations from the literature of VAS in other conditions. For example, in patients with chronic musculoskeletal pain, in a VAS scale of 0 to 10 scores below 3.4 corresponded to mild pain, scores between 3.5 and 7.4 corresponded to moderate pain, and scores above 7.5 corresponded to severe pain. Using such results from other conditions, it is *estimated* that values between 0 and 34 correspond to mild symptoms, scores between 35 and 74 correspond to moderate symptoms, and scores above 75 correspond to severe symptoms.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham+MGX | IPL+MGX
Number analyzed (Participants) | 43 | 39
score on a scale | -25.9 (3.6) | -32.96 (3.97)

4. Other Pre Specified Outcome: Qualitative Assessment of Eyelid Appearance
Description: High resolution photos of the upper and lower eyelids in both eyes
Time Frame: 10 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Meiboscore
Description: The difference in the percentage of area loss of meibomian glands, as evaluated using meibography, between eyes in the study arm and eyes in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percentage of Eyes With Normal Tear Break-Up Time (TBUT)
Description: The difference in the proportion of eyes with normal TBUT (TBUT > 10 sec) at follow-up, between study eyes in the study arm and study eyes in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Percentage of Subjects With Normal Ocular Surface Disease Index (OSDI)
Description: The difference in the proportion of subjects with normal OSDI (OSDI < 23) at FU, between study eyes in the study arm and study eyes in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Incidence of Ocular Adverse Events
Description: The difference in the incidence of ocular adverse events, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Incidence of Non-ocular Adverse Events
Description: The difference in the incidence of non ocular adverse events, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidence of Unanticipated Serious Adverse Events
Description: The difference in the incidence of unanticipated serious adverse events, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Immediate Biomicroscopy
Description: difference in the change of bio-microscopy examinations pre- and post- treatment, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Pain/Discomfort During Intense Pulsed Light (IPL)
Description: The difference in the self-assessment of pain/discomfort during IPL administration, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pain/Discomfort During Meibomian Gland Expression (MGX)
Description: The difference in the self-assessment of pain/discomfort during MGX, between subjects in the study arm and subjects in the control arm
Time Frame: 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Sham+MGX | IPL+MGX
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 9/43 | 4/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sham+MGX (N=43) | IPL+MGX (N=45)
Bronchitis (General disorders) | 1 | 0
Hyperlipidemia (General disorders) | 1 | 0/0
Sinus infection (General disorders) | 2 | 0
worsening of seasonal allergies (General disorders) | 2 | 0
Allergic conjunctivitis (Eye disorders) | 0 | 1
Bacterial conjunctivitis (Eye disorders) | 0 | 1
Conjunctival telangiectasia (Eye disorders) | 1 | 0
Blepharitis (Skin and subcutaneous tissue disorders) | 0 | 1
Chalazion (Skin and subcutaneous tissue disorders) | 1 | 0
Pain (Skin and subcutaneous tissue disorders) | 0 | 1
Stye (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03396913/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT03396913/SAP_001.pdf